CLINICAL TRIAL: NCT06636981
Title: All Trans Retinoic Acid Combined with Toripalimab+Chemotherapy for Locally Advanced Inoperable or Metastatic Triple Negative Breast Cancer：a Multi-center, Multi-cohort Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, MD, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNBC-ATRA-IIT-001
Record Dates: First submitted 2024-09-29; First posted 2024-10-15 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-09

CONDITIONS: Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cohort1: All trans retinoic acid+Toripalimab+Chemotherapy (Experimental)
  Interventions: Drug: Cohort1: ATRA+Toripalimab+chemo
- cohort2: ATRA+Toripalimab+TPC (Experimental)
  Interventions: Drug: Cohort2: ATRA+Toripalimab+TPC

INTERVENTIONS:
Drug: Cohort2: ATRA+Toripalimab+TPC — Receive 200 mg D1 of Toripalimab via intravenous infusion for a course of 21 days; TPC regimen (monoclonal antibody 10mg/kg D1, 8 intravenous infusions, 1 course of treatment every 21 days; Elibulin 1.4mg/m2 D1, 8 intravenous infusions, 1 course of treatment every 21 days; Utideron 40mg/m2 D1-5 intravenous infusions, 1 course of treatment every 21 days; Gemcitabine 1000mg/m2 D1, 8 intravenous infusions, 1 course of treatment every 21 days; Albumin paclitaxel 100 mg/m2 D1, D8, intravenous infusion, 1 course of treatment every 21 days); Capecitabine 1000mg/m2, D1-14, oral, one course of treatment every 21 days); All trans retinoic acid 20 mg bid, orally, D-3-D11, administered continuously for 14 days, stopped for 7 days, with one course of treatment lasting 21 days.
  Arms: cohort2: ATRA+Toripalimab+TPC
Drug: Cohort1: ATRA+Toripalimab+chemo — Receive 200 mg of Toripalimab via D1 intravenous infusion, with 21 days as one course of treatment; Albumin paclitaxel 100 mg/m2, D1, D8, intravenous infusion, one course of treatment for 21 days; All trans retinoic acid 20 mg bid, oral, D-3-D11, continuous administration for 14 days, cessation for 7 days, 21 days is one course of treatment.
  Arms: cohort1: All trans retinoic acid+Toripalimab+Chemotherapy

SUMMARY:
All trans retinoic acid Combined with Toripalimab+Chemotherapy for Locally Advanced inoperable or Metastatic Triple Negative Breast Cancer：a multi-center, multi-cohort phase II trial

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participate and sign a written informed consent form;
2. Age ≥ 18 years old;
3. For locally advanced inoperable or metastatic breast cancer confirmed by histology (according to AJCC 8th edition staging), the histology and pathology clearly showed that ER, PR, Her-2 were negative. If there was metastatic lesion pathology, the metastatic lesion histology and pathology should prevail. The definition of ER and PR negativity is: IHC ER<1%, IHC PR<1%. Her-2 negativity is defined as: immunohistochemical detection of Her-2 (-) or (1+), Her-2 (2+) must undergo FISH testing and the result is negative, Her-2 (-) or (1+) can choose to undergo FISH testing and the result is negative;
4. According to RECIST 1.1 criteria for solid tumor evaluation, there must be at least one measurable lesion;
5. Cohort 1: For locally advanced non operable or metastatic TNBC that has not been previously treated, intravenous chemotherapy and anti-tumor therapy may be used during previous neoadjuvant and/or adjuvant therapy stages, provided that the interval between the end of neoadjuvant and/or adjuvant therapy and the occurrence of recurrence/metastasis is ≥ 12 months; Cohort 2: Local late stage inoperable or metastatic TNBC with previous treatment failures of at least one line or above;
6. All subjects should undergo tumor lesion biopsy during the screening period to obtain sufficient qualified tumor tissue specimens for retrospective biomarker analysis (including PD-L1 expression levels) in their cohort. If subjects are unable to undergo biopsy, they should provide tumor samples or unstained sections (3-5 μm) that have been fixed in formalin and embedded in paraffin (FFPE) closest to the start of the study treatment (up to 24 months) for corresponding biomarker analysis;
7. The main organ function is good, the relevant examination indicators within 14 days before treatment meet the following requirements:

   Without blood transfusion, platelet count ≥ 100 × 10^9/L, hemoglobin ≥ 90g/L, neutrophil count (ANC) ≥ 1.5 × 10^9/L AST and ALT ≤ 2.5 x upper limit of normal (ULN), ≤ 5 x ULN if liver metastasis is present, total bilirubin ≤ 1.5 x ULN, serum creatinine (Cr) ≤ 1.5 ULN, or creatinine clearance rate ≥ 60mL/min (Cockcroft Gault formula)
8. Expected survival period ≥ 3 months;
9. ECOG PS score: 0-1 points;
10. Non surgical sterilization, male patients with women of childbearing age or partners of childbearing age, are required to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill, or condom) during the study treatment period and within 6 months after the end of the study treatment period; Female patients of childbearing age who undergo non-surgical sterilization must have a negative serum HCG test within 72 hours prior to enrollment in the study.

Exclusion Criteria:

1. Individuals who have previously been treated with PD-1 or PD-L1 monoclonal antibodies; Participants in cohort 1 who have previously used albumin paclitaxel;
2. Individuals known to be allergic to any of the drugs in the study;
3. Patients who have hypersensitivity reactions to other vitamin A drugs;
4. History of active autoimmune diseases requiring systemic treatment in the past 2 years (e.g. corticosteroids (dose ≤ 10mg/day, except for prednisone or other effective hormones) or immunosuppressive drugs);
5. Diagnosed with immune deficiency or undergoing systemic steroid therapy (excluding doses ≤ 10mg/day of prednisone or other effective hormones) or any other form of immunosuppressive therapy within 7 days prior to enrollment;
6. There are other known malignant tumors that have progressed or require active treatment in the past 5 years. Excluding malignant tumors that can be treated locally and have already been cured, such as skin basal cell carcinoma, skin squamous cell carcinoma, and cervical cancer in situ;
7. Known to have active central nervous system (CNS) metastases;
8. History of non infectious pneumonia requiring steroid hormone therapy;
9. Active infections require systematic treatment;
10. There are serious uncontrolled hypertension, diabetes and hyperlipidemia;
11. History of II-IV congestive heart failure or myocardial infarction within 6 months prior to enrollment;
12. Individuals who tested positive for HIV during screening;
13. Active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA ≥ 500 IU/ml; hepatitis C reference: HCV antibody positive and HCV copy number>upper limit of normal value);
14. Individuals with other serious acute or chronic physiological or mental problems;
15. Accepting any medication that is prohibited from being used in combination with the investigational drug, unless the medication has been discontinued within 7 days prior to enrollment;
16. Lactating women;
17. Individuals who have participated in clinical trials of other anti-tumor drugs within the past four weeks;
18. Inability to swallow, intestinal obstruction, or other factors that affect medication administration and absorption;
19. Any situation that other researchers consider unsuitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  During the combined therapy, tumor assessment (enhanced CT) is conducted every 3 cycles (6 weeks), and the efficacy is evaluated using the RECIST 1.1 criteria. ORR will be summarized as the proportion of subjects achieving objective tumor responses (complete response or partial response). ORR and its 95% confidence interval will be calculated.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 2 years
  Overall survival (OS) will be defined as time from initiation of therapy to death, or censored at last follow-up date if the Patient is alive and will be calculated based on modified RECIST version 1.1 and iRECIST. Kaplan-Meier methods will be used to estimate OS with 95% CI.
Progression-Free Survival (PFS) | up to 2 years
  Progression free survival (PFS) will be defined as the time from initiation of therapy to the time of RECIST progression or death and will be calculated based on modified RECIST version 1.1 and iRECIST. Kaplan-Meier methods will be used to estimate PFS with 95% CI.
Duration of Response (DOR) | up to 2 years
  DOR is defined as the time from first documented evidence of a CR or PR until progressive disease (PD) or death. DOR for participants who had not progressed or died at the time of analysis will be censored at the date of their last tumor assessment. Per RECIST 1.1
Adverse events | up to 2 years
  Adverse events and toxicity will be assessed according to the NCI-CTCAE 5.0 criteria. Medical review of adverse events and laboratory values will be conducted, and a safety assessment will be completed. Safety assessments will be conducted for all subjects receiving the study drug, with evaluation starting from the date of informed consent signing and continuing until the study concludes or 30 days after drug discontinuation.
Skin adverse reactions | up to 2 years
  Incidence of hand foot syndrome,, maculopapular rash, itching, urticaria, and pigmentation Skin rash and erythema NCI CTCAE level severity Dermatology Quality of Life Questionnaire (DLQI)
Biomarker analysis | up to 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No